CLINICAL TRIAL: NCT01123681
Title: Observational Study of Intubation and Extubation Over 48 Hours Mechanical Ventilation
Brief Title: Intubation and Extubation Over 48 Hours Mechanical Ventilation
Acronym: INDEX48
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Okayama Research Investigator Organizing Network (Network)
Responsible Party: Hiroshi Morimatsu, Okayama University Hospital
Other Study IDs: ORION-INDEX48
Record Dates: First submitted 2010-05-09; First posted 2010-05-14 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Pneumonia, Ventilator-Associated; Critical Illness
Keywords: Respiration, Artificial; Pneumonia, Ventilator-Associated; Critical Illness
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Critical Illness; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ventilator associated pneumonia
  Interventions: Device: Choice of endotracheal tube
- No pneumonia
  Interventions: Device: Choice of endotracheal tube

INTERVENTIONS:
Device: Choice of endotracheal tube — Types of endotracheal tube, normal cuff without sub-glottic aspiration, normal cuff with sub-glottic aspiration, Special cuff with sub-glottic aspiration
  Other Names: Normal cuff without aspiration means Hi-Lo; Normal cuff with aspiration means Hi-Lo Evac; Special cuff with aspiration means Taper Guard

SUMMARY:
The purpose of this study is to determine how often ventilator associated pneumonia happens in the current intensive care units, and how types of endotracheal tube affect its occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years old
* Mechanically ventilated over 48 hours in the ICU

Exclusion Criteria:

* Mask ventilation
* Tracheostomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in an intensive care unit
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence and timing of ventilator associated pneumonia | one month
  From tracheal intubation to ICU duscharge

SECONDARY OUTCOMES:
Ventilator-free days | one month
  During ICU stay
Duration of ICU stay and hospital stay | three months
  From tracheal intubation to ICU or hospital discharge
ICU and hospital mortality | three months
  From tracheal intubation to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Morimatsu, MD, Ph D, Principal Investigator — Okayama University
Locations (6):
- Japan (6):
  - Intensive Care Unit, Himeji Red Cross Hospital, Himeji, Hyōgo
  - Intensive Care Unit, Hiroshima City Hospital, Hiroshima
  - Intensive Crae Unit, Kochi Medical School Hospital, Kochi
  - Intensive Care Unit, Kagawa Rosai Hospital, Marugame
  - Intensive Care Unit, Okayama University Hospital, Okayama
  - Intensive Care Unit, Tsuyama Chuo Hospital, Tsuyama

REFERENCES:
- See also: This is the study homepage written in Japanese. — http://web.me.com/morimatsu1/INDEX_48/Welcome.html